CLINICAL TRIAL: NCT04345042
Title: The Effects of Inhibition of Sternocleidomastoideus Muscle in Patients With Neck Pain
Brief Title: The Inhibition of Sternocleidomastoideus Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Öznur Büyükturan, Assoc. Prof. Öznur BÜYÜKTURAN, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ahi Evran University; Buket Buyukturan (Registry Identifier: Ahi Evran University)
Record Dates: First submitted 2020-04-04; First posted 2020-04-14 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Neck Pain; Massage; Range of Motion
MeSH Terms: conditions — Neck Pain | interventions — Exercise; High-Energy Shock Waves

STUDY DESIGN:
Intervention Model Description: A Single- Blind Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Group (No Intervention): In the first group; the investigators applied the TP such as hot pack, ultrasound, exercise and TENS.
- Second Group (Experimental): In the second group; the investigators applied the classic massage (Swedish Technique) together with TP.
  Interventions: Other: Classic Massage (Swedish Technique)

INTERVENTIONS:
Other: Classic Massage (Swedish Technique) — Classic Massage (Swedish Technique); The massage was applied to the paitents with NP in the second group. Massage procedure included 3 strokes, 3 kneads, and 3 strokes to the upper back and neck area. The application was supported by face cradle and carried out in a semi-horizontal position in which the neck was relaxed. The patient was lying in supine position.
  Other Names: Exercise, transcuteneal electric stimulation, ultrasound, hot pack
  Arms: Second Group

SUMMARY:
Neck pain (NP) is a major public health problem with high prevalence, high cost of health expenditure and loss of productivity.The incidence of NP is increasing among adults and it has been reported to occur in 12-34% of the total population. Exercise programs applied to individuals with NP include craniocervical flexion exercises that focus on the increase in activation of deep cervical flexor muscles and a decrease in the activation of superficial cervical flexors. Falla et al. noted that people with NP also have reduced ability to relax sternocleidomastoideus (SCM) muscle. Although there are many studies indicating that the activation of the SCM muscle should be reduced by activating deep cervical flexors when the literature on NP is examined, there are no studies examining the effect of the inhibition of the SCM muscle.

DETAILED DESCRIPTION:
Patients with NP who were directed to a physiotherapy and rehabilitation program by a specialist physician and meeting the inclusion criteria were included in the study. Criteria for inclusion in the study; NP complaint persists for at least 3 months and is between the ages of 18-55. Exclusion criteria are; Having a history of cervical spine surgery, being included in the physiotherapy and rehabilitation program due to NP in the last 6 months, having a diagnosis of vertebrobasilar artery failure, being diagnosed with cervical stenosis, torticollis, scoliosis, and diagnosing serious pathology such as malignancy, infection and inflammatory disorders.

Outcome measures:

Pain: Visual analog scale (VAS) was used to detect the patients pain intensity. VAS is a simple and common method to evaluate pain intensity. Subjects were instructed to indicate the intensity of their pain by marking a 10-cm line anchored with terms describing the extremes of pain intensity in the last 24 hours. VAS has been shown to be reliable and valid in measuring pain.

Disability: Neck Disability Index (NDI) was applied in order to evaluate how the patient's NP affects their daily life. Total point changes between 0 and 35, with a high score indicating a higher level of disability.

Degree of Cervical Range of Motion (ROM): A universal goniometer was used to assess the Range of Motion of the cervical vertebrae. Cervical flexion, extension, right and left lateral flexion, and right and left rotation movements were measured 3 times in an active manner while the patients were in a comfortable sitting position. The average value of the measurements was recorded as ROM. The pain-free maximum degree of movement for each range was measured in degrees. This method has demonstrated good reliability.

Depressive Symptoms: Participants' level of depression was assessed using Back Depression Inventory that consists of 21 categories with 4 options in each category. Each item has a score between 0 and 3, and total score varies from 0 to 63. Score ranges are interpreted as 0-9 points = minor depression, 10-16 points = mild depression, 17-29 points = moderate depression, and 30-63 points = severe depression.

Kinesiophobia: Tampa scale of kinesiophobia (TSK): The scale was used to assess fear of pain or re-injury that may occur because of any movement. Consisting of 17 items, the scale assesses the parameters of injury/re-injury and fear/avoidance in various activities. Total points may vary between 17 and 68, with a high score indicating a higher level of kinesiophobia.

Evaluation of the static endurance of the neck muscles: Neck extensors and neck flexors endurance test were used to evaluate the static endurance of the neck muscles. Each measurement will be taken 2 times and the best measurement was recorded. Time was given to rest the person for 3 minutes between measurements. The time in which the patient can maintain the position was recorded in seconds.

Neck ﬂexors endurance test; Patients were lying down in the hook lying position with the therapist's hand placed under their head. The patients were then asked to bring their chin closer to their chest in the Chin Tuck position lifting their head about 2.5 cm and to then hold that position. The test was terminated if the patient experienced any pain or fatigue, or if their head touched the therapist's hand. Two measurements were taken and the longest duration was recorded.

Neck extensors endurance test; Patients were lying with their heads bent downwards and their arms resting at their sides. They were asked to approach the edge of the bed so that their head and chest would be hanging from the bed. A sandbag weighing of 2 kg was placed at the back of the neck (between the ears) and the patients were asked to lift their head to the neutral position and then hold it there. The test was terminated in case of any pain or fatigue experienced by the patients, or a 5˚ deterioration in the position of the head. Two measurements were taken and the highest score was recorded.

Randomization: The patients were divided into two groups, according to their age and duration of disease by using matched randomization.

Intervention:

First Group: Traditional physiotherapy (TP) program was applied to patients with NP in the first group. TP program consists of hot-pack, ultrasound, transcutaneal electrical nerve stimulation (TENS) and exercises.

Second Group: The individuals who participated in the second group were applied classical massage and stretching exercises suitable for the SCM muscle together with TP. The treatment program applied to the patient in the first group was applied in the same way. The Classic massage procedure was applied to the SCM for 5 minutes using the Swedish technique. The classic massage was performed by a trained physiotherapist. The procedure included 3 strokes, 3 kneads, and 3 strokes to the upper back and neck area. The application was supported by face cradle and carried out in a semi-horizontal position in which the neck was relaxed. The patient was lying in supine position.

ELIGIBILITY:
Inclusion Criteria:

- Neck pain complaint persists for at least 3 months

Exclusion Criteria:

* History of cervical spine surgery
* Being included in the physiotherapy and rehabilitation program due to neck pain in the last 6 months
* Diagnosis of vertebrobasillar artery failure
* Diagnosed with cervical stenosis, torticollis, scoliosis, and diagnosing serious pathology such as malignancy, infection and inflammatory disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Pain Assessment | 6 weeks
  Visual analog scale was used to detect the patients pain intensity. VAS is a simple and common method to evaluate pain intensity. Subjects were instructed to indicate the intensity of their pain by marking a 10-cm line anchored with terms describing the extremes of pain intensity in the last 24 hours. VAS has been shown to be reliable and valid in measuring pain.
Disability | 6 weeks
  Neck Disability Index (NDI) was applied in order to evaluate how the patient's NP affects their daily life. Total point changes between 0 and 35, with a high score indicating a higher level of disability.

SECONDARY OUTCOMES:
Degree of Cervical Range of Motion | 6 weeks
  A universal goniometer was used to assess the Range of Motion of the cervical vertebrae. Cervical flexion, extension, right and left lateral flexion, and right and left rotation movements were measured 3 times in an active manner while the patients were in a comfortable sitting position. The average value of the measurements was recorded as ROM. The pain-free maximum degree of movement for each range was measured in degrees. This method has demonstrated good reliability.
Depressive Symptoms | 6 weeks
  Participants' level of depression was assessed using Back Depression Inventory that consists of 21 categories with 4 options in each category. Each item has a score between 0 and 3, and total score varies from 0 to 63. Score ranges are interpreted as 0-9 points = minor depression, 10-16 points = mild depression, 17-29 points = moderate depression, and 30-63 points = severe depression.
Kinesiophobia | 6 weeks
  Tampa scale of kinesiophobia was used to assess fear of pain or re-injury that may occur because of any movement. Consisting of 17 items, the scale assesses the parameters of injury/re-injury and fear/avoidance in various activities. Total points may vary between 17 and 68, with a high score indicating a higher level of kinesiophobia.
Evaluation of the static endurance of the neck muscles | 6 weeks
  Neck extensors and neck flexors endurance test were used to evaluate the static endurance of the neck muscles. Each measurement will be taken 2 times and the best measurement was recorded. Time was given to rest the person for 3 minutes between measurements. The time in which the patient can maintain the position was recorded in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Öznur Büyükturan, Principal Investigator — Mr.
Locations (1):
- Ahi Evran University, School of Physical Therapy and Rehablitation, Kırşehir, Others, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sihawong R, Janwantanakul P, Sitthipornvorakul E, Pensri P. Exercise therapy for office workers with nonspecific neck pain: a systematic review. J Manipulative Physiol Ther. 2011 Jan;34(1):62-71. doi: 10.1016/j.jmpt.2010.11.005. PMID 21237409
- [Result] Hogg-Johnson S, van der Velde G, Carroll LJ, Holm LW, Cassidy JD, Guzman J, Cote P, Haldeman S, Ammendolia C, Carragee E, Hurwitz E, Nordin M, Peloso P; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. The burden and determinants of neck pain in the general population: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S39-51. doi: 10.1097/BRS.0b013e31816454c8. PMID 18204398
- [Derived] Buyukturan B, Sas S, Kararti C, Buyukturan O. The effects of combined sternocleidomastoid muscle stretching and massage on pain, disability, endurance, kinesiophobia, and range of motion in individuals with chronic neck pain: A randomized, single-blind study. Musculoskelet Sci Pract. 2021 Oct;55:102417. doi: 10.1016/j.msksp.2021.102417. Epub 2021 Jun 12. PMID 34147954